CLINICAL TRIAL: NCT01228721
Title: Reproducibility of Retinal Nerve Fiber Layer Thickness Measurements Using the Eye Tracker and Retest Function of Spectralis® SD-OCT in Glaucomatous Eyes and Healthy Controls
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Funk Jens, Prof. Dr. Dr., University Hospital Zurich, AUG Augenklinik,
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RNFL-Eyetracker-Foll
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Proton Therapy

INTERVENTIONS:
Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H

SUMMARY:
PURPOSE. To evaluate the impact of self-acting eyetracking and retest software on the reproducibility of retinal nerve fiber layer (RNFL) thickness measurements in glaucoma patients and healthy control subjects using Spectralis® SD-OCT.

METHODS. RNFL thickness was measured in 56 normal and 47 glaucomatous eyes by one operator within one session with a brief rest between measurements. Three measurements were taken with the eye-tracker and retest function, and three were taken without this function, alternating between measurement methods.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* Visual acuity of more or equal to 0.5 Snellen, refractive error less than ±5.00 diopters (D) spheric and ±3.00 D cylindrical and no history of ocular trauma or of any other severe ocular disease (particularly diseases affecting the optic nerve or surgery other than uncomplicated cataract surgery).
* Additional inclusion criteria for the glaucoma group were a diagnosis of primary open angle glaucoma (POAG) or PEX-glaucoma.

Exclusion criteria:

* Exclusion criteria for the control group were history of glaucoma or intraocular pressure beyond 21 mmHg and optic disc cupping of more than 0.6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-01; Study Completion 2010-12

PRIMARY OUTCOMES:
retinal nerve fiber layer thickness measurement

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Langenegger SJ, Funk J, Toteberg-Harms M. Reproducibility of retinal nerve fiber layer thickness measurements using the eye tracker and the retest function of Spectralis SD-OCT in glaucomatous and healthy control eyes. Invest Ophthalmol Vis Sci. 2011 May 18;52(6):3338-44. doi: 10.1167/iovs.10-6611. PMID 21330656